CLINICAL TRIAL: NCT06179056
Title: Anti-microbial Role of Non-antibiotic Agents Against Cutibacterium Acnes in Patients With Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Essam, Lecturer of Dermatology, Zagazig University
Other Study IDs: 10156 IRB
Record Dates: First submitted 2023-11-26; First posted 2023-12-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group
  Interventions: Diagnostic Test: assess the possible role of Salicylic acid, Isotretinoin, and N-acetylcysteine in improving the susceptibility of C. acne for Azithromycin and Doxycycline.

INTERVENTIONS:
Diagnostic Test: assess the possible role of Salicylic acid, Isotretinoin, and N-acetylcysteine in improving the susceptibility of C. acne for Azithromycin and Doxycycline. — Microbiological samples were collected from all patients for:
  1. Isolation of C. acnes
  2. Antibiotic susceptibility testing for C. acnes isolates against the most commonly used antibiotics in the treatment of acne(Azithromycin and Doxycycline) in the presence and absence of Salicylic acid, Isotretinoin, and N-acetylcysteine
  3. Testing biofilm forming ability of C. acnes isolates in the presence and absence of Salicylic acid, Isotretinoin, and N-acetylcysteine

SUMMARY:
* To evaluate and compare the anti-biofilm activity of Salicylic acid, Isotretinoin, and N-acetylcysteine against C. acne .
* To assess the possible role of Salicylic acid, Isotretinoin, and N-acetylcysteine in improving the susceptibility of C. acne for Azithromycin and Doxycycline.

DETAILED DESCRIPTION:
The study was carried out on 24 patients with acne vulgaris. They were recruited from the outpatient clinic of the Dermatology and Venereology and Andrology Department, Zagazig University Hospitals, Egypt.

The degree of severity of lesions was determined by the global acne grading system (GAGS)

Microbiological samples were collected from all patients for:

1. Isolation of C. acnes
2. Antibiotic susceptibility testing for C. acnes isolates aganist the most commonly used antibiotics in treatment of acne(Azithromycin and Doxycycline) in the presence and absence of Salicylic acid, Isotretinoin, and N-acetylcysteine
3. Testing biofilm forming ability of C. acnes isolates in the presence and absence of Salicylic acid, Isotretinoin, and N-acetylcysteine

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients.
* Patients of both sexes.
* Patients with acne vulgaris with different grades

Exclusion Criteria:

* Patients received topical or oral treatment within 6 weeks prior to microbiological sampling

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study was carried out on 48 patients with acne vulgaris
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
inhibition of biofilm formation of c.acne after the use of Salicylic acid, Isotretinoin, and N-acetylcysteine | 6 month
  Biofilm forming ability of P. acnes isolates was adapted from Coenye et al., 2007 and Abbott et al., 2022
  G. The results were obtained according to (Stepanovic et al., 2007); the average OD values were calculated for all tested isolates & negative controls, and the cut-off value (ODc) was detected. It is defined as a 3 standard deviation (SD) above the mean OD of the negative control. The final OD value of a tested strain was expressed as the average OD value of the strain reduced by ODc value; ODc value was calculated for each plate separately. For easier interpretation of the results, strains were divided into the following categories:
  * Non-biofilm producer = OD ≤ODc
  * Strong biofilm producer = 4×ODc <OD
  Growth in the presence of the following agents was tested (all percentages are w/v): 2% salicylic acid, 5% acetylcysteine, and 0.05% isotretinoin
improvement of antibiotic sensitivity of c.acne after the use of Salicylic acid, Isotretinoin, and N-acetylcysteine | 6 month
  All strains were tested for antibiotic susceptibility to azithromycin and doxycycline The minimal inhibitory concentration (MIC) was evaluated by the broth microdilution method according to CLSI (2012). The minimal bactericidal concentration (MBC) was evaluated by using a modified flash microbicide method (Hernandes et al., 2013).
  The MICs of the tested antimicrobial agents were determined by the broth microdilution method according to CLSI (2012) as above in the presence of 2% salicylic acid, 5% acetylcysteine and 0.05% isotretinoin

CONTACTS AND LOCATIONS:
Overall Officials: Reham Essam, Principal Investigator — Zagazig University
Locations (1):
- Reham Essam, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Essam R, Nasr M, Khater MW, Fayez B, Anis N. Anti-microbial impact of non-antibiotic agents; salicylic acid, N-acetylcysteine, and isotretinoin against Cutibacterium acnes in patients with acne vulgaris. Arch Dermatol Res. 2024 Dec 30;317(1):155. doi: 10.1007/s00403-024-03608-7. PMID 39739120